CLINICAL TRIAL: NCT04095611
Title: The Effects of a Modified Muscle Sparing Posterior Technique (SPAIRE) in Hip Hemiarthroplasty for Displaced Intracapsular Fractures on Post-operative Function Compared to a Standard Lateral Approach; a Randomised Controlled Trial
Brief Title: A Modified Muscle Sparing Posterior Technique (SPAIRE) in Hip Hemiarthroplasty for Displaced Intracapsular Fractures.
Acronym: HemiSPAIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS: 258327
Record Dates: First submitted 2019-07-22; First posted 2019-09-19 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Hip Fracture
Keywords: Hemiarthroplasty; Hip fracture; Modified Muscle Sparing Posterior Technique (SPAIRE); Displaced Intracapsular Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The surgeon performing the operation will be aware which treatment the participant is receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPAIRE (Experimental): hemiarthroplasty surgery, the muscle-sparing modification of the posterior approach (SPAIRE).
  Interventions: Procedure: SPAIRE
- LATERAL (Active Comparator): hemiarthroplasty surgery, the standard lateral approach
  Interventions: Procedure: LATERAL

INTERVENTIONS:
Procedure: SPAIRE — To perform the hip surgery called hemiarthroplasty surgeons need to cut through some muscles to expose the hip joint and perform the partial replacement. Currently this often performed using a technique which involves cutting muscles and tendons from the side of the hip and this is called the lateral approach. SPAIRE is a modified technique that accesses the surgical area through a different route.
  Arms: SPAIRE
Procedure: LATERAL — surgery in adults with a displaced intracapsular hip fracture requiring hemiarthroplasty, the standard lateral approach.
  Arms: LATERAL

SUMMARY:
Which technique is best for partial hip replacement?

DETAILED DESCRIPTION:
Aim of study: To compare two ways of performing partial hip replacement to see which one allows patients to mobilise better and gives patients improved function after surgery. The best approach is more likely to allow patients to maintain their independence and return to their own homes after their injury.

Background: When someone breaks their hip they often need a partial hip replacement, also known as hemiarthroplasty. To perform this operation surgeons need to cut through some muscles to expose the hip joint and perform the partial replacement. Currently, clinical guidelines suggest that this operation should be performed using a technique which involves cutting muscles and tendons from the side of the hip. This is called the lateral approach. Alternatively, a newer, modified technique can be used leaving all the major muscles intact and this may cause fewer problems for the patient. There is no research evidence to prove which approach is more beneficial. Patients and carers looking for information about this are likely to become confused by the many opinions of surgeons speaking about preferred techniques. It is therefore important to find out which technique is better for patients, based on research rather than opinion.

Study design: We will randomly allocate patients who agree to be part of the study to have one of the two techniques to partial hip replacement. We can then compare the impact of the two techniques on how well and fully patients mobilise, the level of pain they experience, and the safety of the techniques. We will also contact a number of patients from both treatment groups to discuss their experience of the surgery in more detail.

Patient and public involvement: This study was inspired by patients who said that mobility and speed to regaining independence are the most important outcomes after surgery. Patients and carers will continue to be involved throughout this study, to ensure that the study results are relevant and important to people at risk of breaking their hip.

Dissemination: We will publish the results of this study widely in scientific and other publications accessable to patients and all involved in the treatment of patients with hip fractures. We will work with surgeons, carers and patients to ensure all appropriate networks are aware of the results and that the outcomes are disseminated in an accessible way so that practices can be changed based on the results of this study.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 60+ presenting with an intracapsular hip fractures requiring cemented hip hemiarthroplasty (NICE CG124 2011), and who are resident in the South West of England

Exclusion Criteria:

* Patients that were immobile (unable to walk) before the hip fracture occurred.
* Patients that are not expected to live until post operative day 120 due to chronic illness and are receiving surgery for palliative care.
* Use of femoral stems that are not of a proven stem design, in line with the recommendations set by the NICE clinical guideline on hip fracture management (NICE CG124 2011).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Oxford Hip Score (OHS) | Post operative day 120
  The Oxford Hip Score is a short patient-reported measure of function and pain following hip surgery (Dawson 1996).
  OHS Range: 0-48, with higher scores representing a better outcome

SECONDARY OUTCOMES:
De Morton Mobility Index (DEMMI) | Post operative day 3 and 120
  The De Morton Mobility Index (DEMMI) assessment tool is a functional test that has been validated for acute hip fracture patient rehabilitation (De Morton 2013) and can be used in the early and late post-operative phases. In particular, it measures patient mobility with no reported ceiling effect. It is completed by a research nurse; hence cognitive impairment of the patient need not prevent its use.
  Raw Score Scale: 0-19 DEMMI Score Scale: 0-100 With higher scores indicating a better outcome
Cumulated Ambulation Score (CAS) | Post operative day 3
  The Cumulated Ambulation Score (CAS) is a simple functional tool where patients are assessed daily on their ambulatory capacity by the treating rehabilitation team during the first three post-operative days, having been validated for use with acute hip fracture rehabilitation (Foss et al. 2006) and is intended to be used in the early rehabilitation phase, being applicable to patients of all cognitive levels. It will serve as a secondary outcome of which criteria are readily available in patients' records and will ensure no potential floor effect of evaluation from the DEMMI score.
  CAS Score Scale Range: 0-18, with higher scores indicating better outcomes
Oxford Hip Score (OHS) | Post operative day 3
  The Oxford Hip Score is a short patient-reported measure of function and pain following hip surgery (Dawson 1996).
  OHS Range: 0-48, with higher scores representing a better outcome
Standardised instrument for measuring generic health status: European Quality of Life 5 Dimensions, 5 Levels (EQ-5D-5L) | Post operative day 3 and 120
  A generic utility index capturing 5 dimensions of health-related quality of life (Herdman 2011) 5 dimensions indicating QoL with each dimension scored in a range from 1-5 with higher scores indicating a worse outcome. The scores for each dimension are listed together to indicate a health state, for example '12345'.
  Overall health scale range:0-100 with higher indicating better health
  EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, may be converted into a single index value. Please see website for details.
Numeric pain Rating Scale (NRS) | Post operative day 3 and 120
  Numeric pain Rating Scale (NRS) Participants are asked to indicate their pain in the last 24 hours on a scale from 0-10, with higher scores indicating more pain.
  For details see:
  Dworkin, R. H., Turk, D. C., Farrar, J. T., Haythornthwaite, J. A., Jensen, M. P., Katz, N. P., ... & Carr, D. B. (2005). Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain, 113(1), 9-19.
Analgesia medications used by participants | Post operative day 3 and 120
  Analgesia medication use will be recorded from patient medical notes, with a tick to indicate which (if any) of the following medications are being taken.
  Medications:
  Paracetamol / codeine / ibuprofen or other non-steroidal anti-inflammatory drug (NSAID) / tramadol / morphine / oxycodone / or other
Adverse Events (AE) and Serious Adverse Events (SAE) will be recorded | Throughout study participation, on average 120 days
  AE will be recorded, defined as any negative consequence of care that results in unintended injury or illness that may or may not have been preventable. For example:
  A physical event, A psychological event (e.g., depressed mood). A laboratory event (e.g., elevated blood sugar). An increase in the severity/frequency of a pre-existing symptom or condition
  An AE is considered serious if it poses a threat to the patient's life or functioning.The FDA defines a SAE as any untoward medical occurrence that:
  Results in death, or Is life-threatening (places the patient at risk of death), or Requires or prolongs an existing hospitalization, or Causes persistent or significant disability or incapacity, or Is a birth defect, or Requires medical intervention to prevent one of the above outcomes
  These will include records of surgical complications: categorized as dislocation, nerve injury, vascular injury, periprosthetic fracture, infection, need for re-operation (with reasons).
Length of stay in hospital (acute and super-spell) | Recorded on day of discharge (likely day 4-10 post operation) and through study completion, on average 120 days
  Length of stay in hospital for the acute hospital admission time will be recorded as number of days in hospital. Likely to be between 4 and 10 days. Length of stay will also be recorded for the total Trust stay (super-spell) that includes any time spent at rehabilitation units.
Place of residence | At 3 time points (pre-fracture, on hospital discharge and at POD120). Throughout study participation, on average 120 days
  Participant's place of residence, recorded as:
  * own home,
  * residential/supported living,
  * nursing home or
  * other. These data will be collected from clinical notes to capture location pre-fracture. It will be collected from patient notes indicating the discharge destination, and will be collected at post operative day (POD) 120.
American Society of Anaesthesiologists (ASA) Physical Status Classification | Day of operation
  The ASA measure of physical status of the patient at the time of the operation will be recorded from surgical notes.
  Scale 1-5, with higher indicating worse health status
Qualitative interviews with participants | Post operative day 120
  We will conduct up to 20 semi-structured telephone interviews with patients (10 in each arm) to examine their experience of the impact of surgery and recovery period, including factors such as pain, mobility, function, independence and quality of life. Participants will be sampled from across the hospital sites taking part in the trial. The patient and public involvement group will advise on the design of the interview schedule.
  Interviews will be conducted at POD120
Patient date of birth | Post operative day 3
  Date of birth will be sourced via patient records and checked with patient at POD 3.
Patient gender | Post operative day 3
  Gender will be sourced via patient records and checked with patient at POD 3.
Patient ethnicity | Post operative day 3
  Patient (or consultee if patient cognitively impaired) will be asked to indicate patient ethnicity at POD 3.
Cognition as assessed by surgical team | Day of operation
  Patient level of cognition - (impaired or not impaired) will be obtained from the operation notes.
  Before the operation the surgical team make a clinically informed decision about whether the patient is able to consent to the operation themselves (not impaired) or lacks capacity (impaired) and will need a consultee to consent to surgery on their behalf. The outcome of this assessment (which is derived using the Abbreviated Mental Test (AMT)) is detailed in the patient's medical notes. A broad categorisation of 'impaired' (if patient required a consultee to consent to surgery) or not impaired (if patient was able to consent to surgery themselves) will be derived from the patient's medical notes, and recorded for this study.

CONTACTS AND LOCATIONS:
Overall Officials: John Charity, MD, Study Director — Royal Devon and Exeter NHS Trust
Locations (1):
- Royal Devon and Exeter NHS Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Price A, Ball S, Rhodes S, Wickins R, Gordon E, Aylward A, Cockcroft E, Morgan-Trimmer S, Powell R, Timperley J, Charity J. Effects of a modified muscle sparing posterior technique in hip hemiarthroplasty for displaced intracapsular fractures on postoperative function compared to a standard lateral approach (HemiSPAIRE): protocol for a randomised controlled trial. BMJ Open. 2021 Jun 8;11(6):e045652. doi: 10.1136/bmjopen-2020-045652. PMID 34103316
- [Background] Ball S, McAndrew A, Aylward A, Cockcroft E, Gordon E, Kerridge A, Morgan-Trimmer S, Powell R, Price A, Rhodes S, Timperley AJ, van Horik J, Wickins R, Charity J. Detailed statistical analysis plan for a randomised controlled trial of the effects of a modified muscle sparing posterior technique (SPAIRE) in hip hemiarthroplasty for displaced intracapsular fractures on post-operative function compared to a standard lateral approach: HemiSPAIRE. Trials. 2022 Nov 5;23(1):924. doi: 10.1186/s13063-022-06790-z. PMID 36335403
- [Derived] Ball S, Aylward A, Cockcroft E, Corr A, Gordon E, Kerridge A, McAndrew A, Morgan-Trimmer S, Powell R, Price A, Rhodes S, Timperley AJ, van Horik J, Wickins R, Charity J. Clinical effectiveness of a modified muscle sparing posterior technique compared with a standard lateral approach in hip hemiarthroplasty for displaced intracapsular fractures (HemiSPAIRE): a multicenter, parallel-group, randomized controlled trial. BMJ Surg Interv Health Technol. 2024 Jun 17;6(1):e000251. doi: 10.1136/bmjsit-2023-000251. eCollection 2024. PMID 38895600